CLINICAL TRIAL: NCT03617198
Title: A Pilot Study of T Cells Genetically Modified by Zinc Finger Nucleases SB-728mR and CD4 Chimeric Antigen Receptor in HIV-infected Subjects
Brief Title: CD4 CAR+ ZFN-modified T Cells in HIV Therapy
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 831464
Record Dates: First submitted 2018-07-09; First posted 2018-08-06 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Experimental): Cohort 1 subjects will begin treatment interruption approximately 24 hours after they receive the modified T-cells. All other study procedures are the same as Cohort 2.
  Interventions: Biological: CD4 CAR+CCR5 ZFN T-cells
- Cohort 2 (Experimental): Cohort 2 subjects will begin treatment interruption approximately 8 weeks after they receive the modified T-cells. All other study procedures are the same as Cohort 1.
  Interventions: Biological: CD4 CAR+CCR5 ZFN T-cells

INTERVENTIONS:
Biological: CD4 CAR+CCR5 ZFN T-cells — A dual cohort, open-label, randomized study of the safety and tolerability of a single infusion of autologous T cells genetically modified to express a CD4 chimeric antigen receptor while also having zinc finger nuclease-mediated disruption of the CCR5 gene

SUMMARY:
This research study is being carried out to study a new way to possibly treat HIV. As part of this study, doctors will take some of your own white blood cells, called T-cells, and modify them so that they can identify and target your HIV cells. The purpose of the study is to evaluate the safety of these modified T cells and determine whether they have any effect on HIV infection.

DETAILED DESCRIPTION:
Step 1:

Subject is screened, undergoes leukaphereses, and optional rectal biopsy, and safety evaluations before dosing. The University of Pennsylvania manufactures the study product.

Step 2:

Subjects receive a single infusion of 0.5-1x10(10) CD4 CAR+CCR5 ZFN modified T cells. Cohort 2 participants undergo a mini-leukapheresis and optional rectal biopsy at the end of step 2.

The duration of Step 2 will be:

* Cohort 1: 1 day
* Cohort 2: 8 weeks

Step 3:

All subjects will participate in a 16 week analytical treatment interruption (ATI). ATI will be less than 16 weeks if patient's viral load is sustained >100,000 or CD4 count <350 or less than 50% of baseline. At the end of step 3 all participants will undergo mini-leukapheresis and optional rectal biopsy.

Step 4:

Participants who have HIV viral loads ≤1000 copies/ml will continue in an extension of the analytical treatment interruption until viral load is sustained >100,000 or CD4 count <350 or less than 50% of baseline.

Step 5:

Reinitiation of antiretroviral therapy with monthly visits until the HIV RNA is below the limit of quantification. All participants undergo a mini-leukapheresis and optional rectal biopsy at the end of the step 5.

Step 6 (Secondary Follow-up):

All subjects will be followed for safety for up to 5 years post-infusion.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* Clinically stable on first or second HAART regimen
* Screening CD4+ T cell count of ≥450 cells/mm3 within 30 days of enrollment; and a documented CD4 nadir of not lower than 200 cells/mm3
* Screening HIV-1 RNA that is ≤50 copies/mL within 30 days prior to enrollment
* HIV-1 RNA ≤50 copies/mL for at least 24 weeks prior to enrollment
* Adequate venous access and no other contraindications for leukapheresis
* Laboratory values within certain parameters, obtained within 30 days prior to enrollment
* Willing to comply with study-mandated evaluations
* Male or female, 18 years of age or older
* Ability and willingness to provide informed consent
* Karnofsky Performance Score of 70 or higher
* Negative HBsAg (hepatitis B) within 6 months prior to enrollment
* Negative HCV (hepatitis C) serology, or if positive, negative HCV RNA within 6 months prior to enrollment
* Have a recorded viral load set point prior to starting antiretroviral therapy

Exclusion Criteria:

* Acute or chronic hepatitis B or hepatitis C infection
* Current or prior AIDS diagnosis
* History of cancer or malignancy, with the exception of successfully treated basal cell or squamous cell carcinoma of the skin
* History or any features on physical examination indicative of active or unstable cardiac disease or hemodynamic instability (subjects with a history of cardiac disease may participate with a physician's approval)
* History or any features of physical examination indicative of bleeding diathesis
* Have been previously treated with any HIV experimental vaccine within 6 months prior to screening, or any previous gene therapy using an integrating vector (subjects treated with placebo in an HIV vaccine study will not be excluded if documentation that they received placebo is provided)
* Use of chronic systemic corticosteroids, hydroxyurea, or immunomodulating agents within 30 days prior to enrollment (recent or current use of inhaled steroids is not exclusionary)
* Breast-feeding, pregnant, or unwilling to use acceptable methods of birth control
* Anticipated use of aspirin, dipyridamole, warfarin, or any other medication that is likely to affect platelet function or other aspects of blood coagulation during the 2 week period prior to leukapheresis
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements
* Serious illness requiring systemic treatment and/or hospitalization within 30 days prior to the study screening visit
* Receipt of vaccination within 30 days prior to study screening visit
* Have an allergy to hypersensitivity to study product components (human serum albumin, DMSO and Dextran 40)
* Currently taking a non-nucleoside reverse transcriptase inhibitor (NNRTI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with treatment related adverse events. | After subjects have received infusion and up to 5 years from Day 0 infusion.

SECONDARY OUTCOMES:
Compare the percentage of enriched modified CD4 CAR+ CCR5 ZFN cells and their subsets. | 2 weeks post infusion, prior to prior to analytical treatment interruption (ATI), 6-9 months post infusion.
Compare the change in CD4 count. | Baseline, week 2 post infusion, prior to ATI, weeks 8, 12, 16 of ATI.
Compare viral set point log 10 HIV RNA level. | Baseline and 6-9 months post infusion
Percentage of cells producing cytokines in response to HIV antigen/peptide as assessed by flow cytometry | Baseline and 6-9 months post infusion
Size of latent HIV reservoir as assessed by quantification of integrated copies of replication competent HIV | Baseline, pre-treatment interruption, prior to ART reinitiation, 6-9 months post infusion, and end of primary follow up (8-12 months)
Sequence of HIV envelope genes and coreceptor usage in breakthrough HIV infections | Baseline through 1 year.
Number of participants who control HIV replication that have similar gene expression patterns as determined by RNA quantification | Baseline through 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Tebas, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No